CLINICAL TRIAL: NCT01473394
Title: A Double-blind, Placebo-controlled, Fixed-dose Study of Vilazodone in Patients With Major Depressive Disorder
Brief Title: Safety, Efficacy, and Tolerability of Vilazodone in Major Depressive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VLZ-MD-03
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Results first posted 2014-04-03 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-02

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Vilazodone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose-matched placebo (Placebo Comparator): Participants received dose-matched placebo orally once daily for 9 weeks.
  Interventions: Drug: Dose-matched placebo
- Vilazodone (Experimental): Participants received vilazodone orally once daily for 9 weeks, as follows: Week 1, 10 mg once a day; Week 2, 20 mg once a day; Weeks 3 to 8, 40 mg once a day; and Week 9 (down-taper period), 20 mg once a day for 4 days, then 10 mg once a day for 3 days.
  Interventions: Drug: Vilazodone

INTERVENTIONS:
Drug: Dose-matched placebo — Dose-matched placebo was supplied as tablets.
  Arms: Dose-matched placebo
Drug: Vilazodone — Vilazodone was supplied as tablets.
  Other Names: Viibryd
  Arms: Vilazodone

SUMMARY:
The purpose of this study was to further characterize the efficacy, safety, and tolerability of a single fixed dose level of vilazodone compared to placebo in patients with major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18-70 years of age.
* Currently meet the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV-TR) criteria for Major Depressive Disorder.
* The patient's current major depressive episode must be at least 8 weeks and no longer than 12 months in duration.

Exclusion Criteria:

* Women who are pregnant, women who will be breastfeeding during the study, and women of childbearing potential who are not practicing a reliable method of birth control.
* Patients with a history of meeting DSM-IV-TR criteria for any:

  * manic, hypomanic or mixed episode, including bipolar disorder and substance-induced manic, hypomanic, or mixed episode;
  * any depressive episode with psychotic or catatonic features;
  * panic disorder with or without agoraphobia;
  * obsessive-compulsive disorder;
  * schizophrenia, schizoaffective, or other psychotic disorder;
  * bulimia or anorexia nervosa;
  * presence of borderline personality disorder or antisocial personality disorder;
  * mental retardation, dementia, amnesia, or other cognitive disorders;
  * patients who are considered a suicide risk.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2011-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Gommoll, MS, Study Director — Forest Laboratories
Locations (14):
- United States (14):
  - Forest Investigative Site 009, Beverly Hills, California
  - Forest Investigative Site 003, Encino, California
  - Forest Investigative Site 010, New Port Beach, California
  - Forest Investigative Site 005, Jacksonville, Florida
  - Forest Investigative Site 004, Orlando, Florida
  - Forest Investigative Site 012, Atlanta, Georgia
  - Forest Investigative Site 001, Baltimore, Maryland
  - Forest Investigative Site 002, Dayton, Ohio
  - Forest Investigative Site 011, Philadelphia, Pennsylvania
  - Forest Investigative Site 015, Lincoln, Rhode Island
  - Forest Investigative Site 008, Memphis, Tennessee
  - Forest Investigative Site 016, San Antonio, Texas
  - Forest Investigative Site 006, Bellevue, Washington
  - Forest Investigative Site 013, Seattle, Washington

REFERENCES:
- [Derived] Kornstein S, Chang CT, Gommoll CP, Edwards J. Vilazodone efficacy in subgroups of patients with major depressive disorder: a post-hoc analysis of four randomized, double-blind, placebo-controlled trials. Int Clin Psychopharmacol. 2018 Jul;33(4):217-223. doi: 10.1097/YIC.0000000000000217. PMID 29608461
- [Derived] Croft HA, Pomara N, Gommoll C, Chen D, Nunez R, Mathews M. Efficacy and safety of vilazodone in major depressive disorder: a randomized, double-blind, placebo-controlled trial. J Clin Psychiatry. 2014 Nov;75(11):e1291-8. doi: 10.4088/JCP.14m08992. PMID 25470094
- [Derived] Citrome L, Gommoll CP, Tang X, Nunez R, Mathews M. Evaluating the efficacy of vilazodone in achieving remission in patients with major depressive disorder: post-hoc analyses of a phase IV trial. Int Clin Psychopharmacol. 2015 Mar;30(2):75-81. doi: 10.1097/YIC.0000000000000056. PMID 25396353

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dose-matched Placebo | Vilazodone
Started | 253 | 255
Completed | 208 | 212
Not Completed | 45 | 43
Not completed — Adverse Event | 13 | 16
Not completed — Insufficient Therapeutic Response | 4 | 1
Not completed — Protocol Violation | 7 | 5
Not completed — Withdrew Consent | 12 | 10
Not completed — Lost to Follow-up | 9 | 11

BASELINE CHARACTERISTICS:
Population: Safety population: All randomized participants who received at least 1 dose of double-blind investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose-matched Placebo | Vilazodone | Total
Number analyzed (Participants) | 253 | 255 | 508
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.1 (13.2) | 39.3 (12.8) | 40.2 (13.0)
Age, Customized [Number; unit: Participants]
  < 20 | 7 | 6 | 13
  ≥ 20-29 | 53 | 68 | 121
  ≥ 30-39 | 54 | 56 | 110
  ≥ 40-49 | 67 | 62 | 129
  ≥ 50-59 | 48 | 44 | 92
  ≥ 60 | 24 | 19 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 131 | 273
  Male | 111 | 124 | 235
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 42 | 75
  Not Hispanic or Latino | 220 | 213 | 433
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 168 | 174 | 342
  Black or African American | 70 | 52 | 122
  Asian | 7 | 14 | 21
  American Indian or Alaska Native | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Other | 7 | 11 | 18
Weight [Mean (Standard Deviation); unit: kg] | 84.68 (17.84) | 82.89 (18.39) | 83.78 (18.12)
Height [Mean (Standard Deviation); unit: cm] | 170.15 (9.12) | 170.32 (9.60) | 170.23 (9.36)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 29.08 (5.50) | 28.41 (5.47) | 28.75 (5.49)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score at Week 8
Description: The MADRS is a clinician-rated scale for assessing depressive symptomatology that had occurred in participants during the week preceding each interview. Patients were rated on 10 items to assess feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and lack of interest. Each item was scored on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). The total score was the sum of the scores on the 10 items and ranged from 0 to 60. A higher score indicated more depressive symptomatology. A negative change score indicated improvement.
Time Frame: Baseline to Week 8
Population: Intent-to-treat population: All randomized participants who received at least 1 dose of double-blind investigational product and who had a Baseline and at least 1 post-baseline assessment of the MADRS total score.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Dose-matched Placebo | Vilazodone
Number analyzed (Participants) | 252 | 253
Units on a scale | -11.0 (0.65) | -16.1 (0.64)
Statistical Analysis 1: Comparison: Dose-matched Placebo vs Vilazodone; Test type: Superiority or Other; p < 0.00001, Mixed-effects model for repeated measure; Least square mean difference = -5.117, 95% CI 2-sided [-6.886 to -3.347]

2. Secondary Outcome: Change From Baseline in Clinical Global Impressions-Severity (CGI-S) Score at Week 8
Description: The CGI-S is a clinician-rated scale for assessing the severity of the participant's current state of mental illness compared with a patient population with major depressive disorder. The clinician responded to the following question "Considering your total clinical experience with this population, how mentally ill is the participant at this time?" on a 7-point scale: 1=normal, not at all ill; 2=borderline ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients. The scale ranges from 1 to 7. A higher score indicates more severe mental illness. A negative change score indicates improvement.
Time Frame: Baseline to Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Dose-matched Placebo | Vilazodone
Number analyzed (Participants) | 252 | 253
Units on a scale | -1.2 (0.08) | -1.8 (0.08)
Statistical Analysis 1: Comparison: Dose-matched Placebo vs Vilazodone; Test type: Superiority or Other; p < 0.00001, Mixed-effects model for repeated measure; Least square mean difference = -0.622, 95% CI 2-sided [-0.845 to -0.399]

3. Secondary Outcome: Percentage of Participants With a Montgomery-Åsberg Depression Rating Scale (MADRS) Sustained Response Rate
Description: The MADRS Sustained response rate is defined as a MÅDRS total score ≤ 12 for at least the last 2 consecutive visits during the double-blind treatment period.
Time Frame: Baseline to Week 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dose-matched Placebo | Vilazodone
Number analyzed (Participants) | 252 | 253
Percentage of participants | 17.1 [12.4 to 21.7] | 27.3 [21.8 to 32.8]
Statistical Analysis 1: Comparison: Dose-matched Placebo vs Vilazodone; Test type: Superiority or Other; p = 0.0047, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 10.2, 95% CI 2-sided [3.0 to 17.4] — The Mean Difference (Final Values), as well as the 95% Confidence Interval, are in units of percentage

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the time the participant signs the informed consent form until 30 days after the last dose of treatment (up to 13 weeks).
Description: Safety population: All randomized participants who received at least 1 dose of double-blind investigational product. The Severe Adverse Event data presented here is for the safety population. The Other Adverse Event data presented here is for the safety population during the 8 week double-blind treatment period.
Arm/Group | Dose-matched Placebo | Vilazodone
Serious Adverse Events (participants affected / at risk) | 2/253 | 3/255
Other Adverse Events (participants affected / at risk) | 78/253 | 149/255
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose-matched Placebo (N=253) | Vilazodone (N=255)
Non-cardiac chest pain (General disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose-matched Placebo (N=253) | Vilazodone (N=255)
Diarrhoea (Gastrointestinal disorders) | 26 | 83
Nausea (Gastrointestinal disorders) | 21 | 63
Headache (Nervous system disorders) | 26 | 24
Dizziness (Nervous system disorders) | 7 | 18
Insomnia (Psychiatric disorders) | 3 | 15
Upper respiratory tract infection (Infections and infestations) | 14 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study.

Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.